CLINICAL TRIAL: NCT02859649
Title: Gestural Short Term and Working Memory Task
Acronym: GeSTWoM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P/2016/283
Record Dates: First submitted 2016-04-14; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Neuropsychology; Gesture
Keywords: working memory; short term memory; gesture
MeSH Terms: conditions — Gestures | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Behavioral: neuropsychological test

INTERVENTIONS:
Behavioral: neuropsychological test — neuropsychological test

SUMMARY:
According to the working memory model, which accounts for the organisation of working memory, the processing of non-meaningful gestures is not clear. Some authors suggest that working memory for non-meaningful gestures has the same characteristics as the phonological loop, made up of a phonological store and of a revival process (articulatory rehearsal). These characteristics are evidenced in memory span tasks, memory span which is itself determined by the duration of the memory trace and the time required to refresh the trace by subvocal rehearsal.

The investigators therefore aim to set up a gestural working memory task, which is specific, simple and reproducible, in the manner of verbal and visuospatial span tasks. It will first be an exploratory and descriptive study with healthy subjects.

DETAILED DESCRIPTION:
In the first instance, each subject performs the gestural working memory test. The test is based on the model of verbal or visuospatial working memory tests. Video clips that display the movement of two, then three, then four different fingers are shown to the subject, who must then reproduce them. There are nine different sub-tests: forward span and backward span for both hands then for each hand, i.e. six sub-tests, in addition to three sub-tests with concomitant interference tasks (verbal, gestural or both). Each sub-test comes to an end when the subject fails both attempts of the same item. The entire test takes approximately 30 minutes.

A questionnaire is then handed to the subject: the subject provides their full name, date of birth, profession, education level (number of years of study post compulsory education), laterality, as well as potential professional or leisure activities that might involve fine finger movement. They also complete the Edinburgh Handedness Inventory assessment.

In order to correlate this new test with other validated tasks, each subject is then required to perform a verbal and visuospatial working memory task: the digit span test and then the spatial memory test, which last approximately 10 minutes.

The entire protocol lasts approximately 45 minutes per subject. The data is then anonymized and processed confidentially.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers
* 18/50 years old
* they must speak fluent French and give their informed consent

Exclusion Criteria:

* neurological or psychiatric disorder
* uncorrected visual or hearing loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Gestural span | 1 day
  Measure and description of the gestural span during the tests of short-term memory and gestural working memory, and correlation with the verbal and visuo-spatial spans.

CONTACTS AND LOCATIONS:
Locations (1):
- Eloi Magnin, Besançon, France

REFERENCES:
- [Background] Baddeley A. The episodic buffer: a new component of working memory? Trends Cogn Sci. 2000 Nov 1;4(11):417-423. doi: 10.1016/s1364-6613(00)01538-2. PMID 11058819
- [Background] Baddeley AD, Allen RJ, Hitch GJ. Binding in visual working memory: the role of the episodic buffer. Neuropsychologia. 2011 May;49(6):1393-400. doi: 10.1016/j.neuropsychologia.2010.12.042. Epub 2011 Jan 20. PMID 21256143
- [Background] Wilson M, Fox G. Working memory for language is not special: evidence for an articulatory loop for novel stimuli. Psychon Bull Rev. 2007 Jun;14(3):470-3. doi: 10.3758/bf03194091. PMID 17874590
- [Background] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997
- [Background] Cowan N. The magical number 4 in short-term memory: a reconsideration of mental storage capacity. Behav Brain Sci. 2001 Feb;24(1):87-114; discussion 114-85. doi: 10.1017/s0140525x01003922. PMID 11515286
- [Background] CONRAD R, HULL AJ. INFORMATION, ACOUSTIC CONFUSION AND MEMORY SPAN. Br J Psychol. 1964 Nov;55:429-32. doi: 10.1111/j.2044-8295.1964.tb00928.x. No abstract available. PMID 14237884